CLINICAL TRIAL: NCT03598972
Title: the Effect of Prenatal Vitamins on the Children Teeth: Elementary Analysis
Brief Title: the Effect of Prenatal Vitamins on the Tooth Structure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina mounir elkady, assistant lecturer, Cairo University
Other Study IDs: 57890
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control: teeth of children of non vitamin taking mother
  Interventions: Other: intervention
- intervention: children teeth of vitamin taking mother
  Interventions: Other: intervention

INTERVENTIONS:
Other: intervention — elementary analysis

SUMMARY:
the effect of mother prenatal care on the teeth of the newborn children, if it affect the tooth structure or not

DETAILED DESCRIPTION:
teeth lost due to normal shedding will be collected,it will be classified into mother that take pregnancy vitamins and mother that doesn't take pregnancy vitamins, the female will be from the same population and from the same city to make sure that the environmental condition are almost the same .teeth will be subjected to elementary analysis to determine the different ratio of different component and if there is any change between the two group

ELIGIBILITY:
Inclusion Criteria teeth lost due to normal shedding sound teeth with non hereditary conditions normal children mother that don not suffer from chronic illness ex: diabetes

Exclusion Criteria:

* teeth extracted due to caries or trauma teeth with hereditary anomalies ex: hypoplasia

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: healthy children within the normal period of teeth shedding
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-06-15 (Estimated); Primary Completion 2021-07-15 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
the different teeth minerals and component | 3months
  analysis of exofilated teeth mineral ratio

SECONDARY OUTCOMES:
caries index of chlidren | 3 months
  dmf index for every patient to count the total missed and decayed teeth

IPD SHARING:
Plan to Share IPD: Undecided